CLINICAL TRIAL: NCT01001533
Title: A Pilot Study to Assess the Ability of Non-invasive Bio-impedance Cardiac Monitoring to Detect and Trend Hemodynamic Variables During Dexmedetomidine (DEX) Sedation in Children for Radiology Procedures
Brief Title: Assess the Ability of Electrical Cardiometry to Trend Hemodynamic Variables During Dexmedetomidine Sedation
Acronym: DEX-CO
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jackson Wong, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 09-03-0130
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2011-06

CONDITIONS: Cardiac Output; Sedation
Keywords: Electrical Cardiometry; Dexmedetomidine; ICON; bio-impedance; cardiac monitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children sedated by DEX: All pediatric patients (1 month to 18 years of age) eligible for Radiology Sedation Service for CT scan and Nuclear Medicine Scan procedure.

SUMMARY:
The aim of the study is to investigate the use of a new FDA-approved non-invasive bio-impedance cardiac monitor, ICON, to detect hemodynamic effects during sedation in children undergoing radiology procedures. The purpose of the study is to determine the ability of the ICON monitor to identify the anticipated and documented hemodynamic changes in children which occur in response to Dexmedetomidine sedation. The investigators postulate that if the ICON device can trend hemodynamic changes, if any, during dexmedetomidine (DEX) sedation in children the investigators can delineate changes in cardiac output, stroke volume, and systemic vascular resistance associated with observed changes in heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (1 month to 18 years of age)
* Eligible for Radiology Sedation Service for CT scan and Nuclear Medicine
* Scan procedure

Exclusion Criteria:

* Pacemakers and Vagus Nerve Stimulator
* Mitral or Aorta Valve Dysfunction
* Dextrocardia
* Second or Third degree heart block
* Current diagnosis of Cardiac, Pulmonary, Hepatic or Renal Failure
* Current diagnosis of pulmonary masses/tumor/pleural effusions/pneumonia/edema
* Pericardial effusion
* Concomitant use of hypertension medications including ACE inhibitors, beta receptor and calcium channel blockers.
* Large Implanted Metallic Devices (including orthodontic braces, spine rods, plates and screws)
* Allergy to device electrodes

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients (1 month to 18 years of age) eligible for Radiology Sedation Service for CT scan and Nuclear Medicine Scan procedure who agrees to participate in the study will have their vital signs and ICON measurements recorded continuously pre-sedation, during sedation and through recovery until discharge.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary aim is to ascertain if a decrease in heart rate (HR) with intravenous (IV) DEX is associated with a change in trend of cardiac output (CO) as measured by the ICON device. | pre-, during, and post sedation

SECONDARY OUTCOMES:
To determine the cardiac parameters provided by the ICON device during changes in blood pressure. | pre-, during and post sedation

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Wong, MD, Principal Investigator — Children Hospital Boston
Locations (1):
- Children Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wong J, Steil GM, Curtis M, Papas A, Zurakowski D, Mason KP. Cardiovascular effects of dexmedetomidine sedation in children. Anesth Analg. 2012 Jan;114(1):193-9. doi: 10.1213/ANE.0b013e3182326d5a. Epub 2011 Sep 29. PMID 21965374